CLINICAL TRIAL: NCT02260115
Title: A Randomized, Controlled, Subject and Reviewer-Blinded, Multi-Centre Study To Assess The Safety and Manageability Of LABS™ In Women Undergoing Gynaecologic Laparoscopic Surgery Followed By Second Look Laparoscopy
Brief Title: A Randomized Multi-centre Study to Assess the Safety and Manageability of a Laparoscopic Adhesion Barrier in Women Undergoing Gynecologic Laparoscopic Surgery Followed by Second Look Laparoscopy
Acronym: LABS-1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Actamax Surgical Materials LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ABS-01EU-2013; 95.10 - 5660 - 7811 (Other: Competent Authority)
Record Dates: First submitted 2014-10-01; First posted 2014-10-09 (Estimated); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Tissue Adhesions
MeSH Terms: conditions — Tissue Adhesions

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LABS™ (Experimental): hydrogel sprayed laparoscopically over all pelvic areas of surgical trauma
  Interventions: Device: LABS™
- Surgical Control (Sham Comparator): Laproscopic Surgery Only
  Interventions: Procedure: Surgical Control

INTERVENTIONS:
Device: LABS™ — hydrogel sprayed laparoscopically over all pelvic areas of surgical trauma
  Arms: LABS™
Procedure: Surgical Control — Surgery only
  Arms: Surgical Control

SUMMARY:
The purpose of this study is to obtain data on the safety and manageability of applying LABS™ to the uterus and other areas of surgical trauma in the pelvis and abdomen following laparoscopic gynaecologic surgery. In addition, performance data following a clinical indicated second look laparoscopy will be collected for the purpose of determining sample size predictions for future trials.

DETAILED DESCRIPTION:
Women undergoing laparoscopic uterine myomectomy, adhesiolysis, treatment of endometriosis or ovarian cystectomy with associated adhesions and/or endometriosis, and planned, clinically indicated second look laparoscopy within 4-12 weeks will be enrolled into one of two sub studies in which the major component of the surgery (as determined by the surgeon) was due to:

1. Myomectomy Or
2. Other Gynaecology Pathology (repeat myomectomy, adhesiolysis, and/or treatment of endometriosis, ovarian cystectomy with associated adhesions or endometriotic pathology, removal of adenomyoma without myomectomy.

The myomectomy sub study will include two arms:

1. Pure Myomectomy -myomectomy with no endometriosis and no adhesions/few filmy uterine adhesions - blunt dissection only
2. Hybrid Myomectomy - myomectomy with (+/-) adhesions and/or (+/-) endometriosis and/or (+/-) adenomyomectomy Patients in each sub study (1 or 2) and each arm of the myomectomy study (a or b) will be randomized to receive LABS™ following their laparoscopic surgery or current standard of care: surgery only control. All patients will be blinded to their treatment status until study completion.

Sub study and sub-group allocation as well as randomisation will occur once the initial laparoscopy is completed but before removal of the laparoscope. Myomectomy patients randomized to receive LABS™ will then have the device sprayed to the entire surface of the uterus and other areas of surgical trauma. In all treated patients all sites of surgical trauma should be completely covered with LABS™ allowing a sprayed margin of at least 3 cm around the operated or traumatised site.

Patients receiving LABS™ will be compared to patients who have had the current standard of care: surgery alone. In addition to an overall comparison, they will be compared to patients in the same sub study (1 or 2) and same arm of the myomectomy study (1a or 1b).

The first two patients entered by each operating surgeon will be allocated to LABS™ and assessed for the application of LABS™. They will not be counted as fully evaluable randomized patients. These patients will be sequentially assigned and evaluated. With confirmatory evaluation of and application of LABS™ on the first patient, the surgeon will be advised to assign the second. With the same confirmatory evaluation on the second patient and both patients discharged from hospital the surgeon will be permitted to proceed with the study and randomise patients.

Both the initial laparoscopic procedure and the clinically indicated second look laparoscopy will be video recorded to allow for a blinded evaluation of LABS™ application and a separate blinded evaluation of adhesions and other pathology in all patients - treated and controls. This evaluation will be cross checked with the operating surgeon's own evaluations and reconciled according to a specified protocol.

Where, during initial surgery, a second look laparoscopy is no longer considered clinically indicated but the surgeon randomizes the patient, they will be followed for safety evaluations only.

ELIGIBILITY:
PREOPERATIVE INCLUSION

Preoperatively the patient must:

* understand and be able to follow the requirements of the protocol including signing and dating an Ethics Committee approved Informed Consent prior to undergoing any protocol related procedures
* be a premenopausal female who is > 18 and < 46 years old
* be thought to have gynaecologic pathology requiring laparoscopic surgery - including uterine fibroids (including those with only anterior fibroid or repeat myomectomy/previous uterine artery embolization for fibroid), adhesions, and/or endometriosis with or without associated pathology such as ovarian cysts
* wish to retain her fertility
* and thus be considered to clinically benefit from a second-look laparoscopic procedure;
* have a willingness to undergo a second-look surgical procedure if clinically indicated
* have a negative pregnancy test within 5 days of surgery
* agree to avoid pregnancy using adequate forms of contraception through the time of performance of second-look laparoscopy (oral contraceptive pill, condom, no sexual intercourse), and if the patient is undergoing myomectomy that she is aware that it is good advice to avoid pregnancy for a 12 week period to allow healing of the uterine scar before becoming pregnant
* be in good health including an ASA (American Society of Anaesthesiologists) score of 2 or less
* following physical and medical assessment have no clinically significant or relevant abnormalities.

PREOPERATIVE EXCLUSION

Preoperatively a patient must not:

* be unable to give their own written informed consent,
* have completed her family planning with no desire to maintain fertility,
* be considered to have no potential clinical benefit from a second look laparoscopy,
* be breastfeeding,
* be within 6 weeks post-partum
* have received or is expected to receive another anti-adhesive treatment within 30 days prior to enrolment or during enrolment up to adhesion evaluation at second look laparoscopy,
* be currently enrolled in another clinical study or has been in another study within the last 30 days,
* have received or is expected to receive any other investigational product or technique within 30 days prior to or during enrolment,
* have had cancer within 5 years of the initial surgery with the exception of basal cell carcinoma,
* have known allergy to dextran, PEG, or FD&C Blue #1,
* be scheduled to undergo concomitant non-gynaecological surgery,
* be currently pregnant (including ectopic pregnancy),
* have received GNRH agonist/antagonist, Depo Provera, danocrine, ulipristal acetate or similar treatment (except oral contraceptives - and including progesterone only) in the 4 weeks prior to study,
* on pre-operative imaging have
* Largest fibroid < 2 cms
* Or largest fibroid > 10 cms diameter intramural
* Or more than 5 large fibroids (large = >8 cms diameter)
* And/or adenomyoma >10cm identified
* have a history where it is expected that complete adhesiolysis will not be possible,
* preoperatively have clinically significant abnormal blood results including:
* SGOT, SGPT and/or bilirubin > 20% above the upper range of normal and/or
* BUN and creatinine > 30% above the upper range of normal,
* have clinically relevant hemochromatosis, hepatic, renal, autoimmune, lymphatic, haematological or coagulation disorders,
* have insulin dependent diabetes mellitus,
* be receiving concurrent systemic corticosteroids, antineoplastic agents and/or radiation therapy,
* have had previous radiation therapy,
* have active pelvic or abdominal infection, or other active infection with fever >38°C.

INTRAOPERATIVE INCLUSION

During surgery the patient must have:

• treatment of uterine fibroids, endometriosis, and or adhesions, with or without associated pathology such as ovarian cysts, and meets all intraoperative inclusion/exclusion criteria prior to randomisation, including that a SLL is clinically indicated

Additionally for the myomectomy sub study, during surgery it must be confirmed that:

* the patient underwent a laparoscopic myomectomy with at least (1) posterior uterine serosal incision of > 3 cm in length
* that the major portion of the procedure (in the opinion of the surgeon) was related to myomectomy
* that the patient meets all intraoperative inclusion/exclusion criteria prior to randomisation.

and

• at the completion of the procedure, prior to randomisation, the surgeon continues to believe that the patient will clinically benefit from second- look laparoscopy.

INTRAOPERATIVE EXCLUSION

Intraoperatively a patient must not:

* have cancer detected at surgery,
* be pregnant, including ectopic pregnancy,
* have a non-gynaecological surgical procedure or entry into the bowel, bladder, or ureter,
* have a hysterectomy or other gynaecological procedure that would render the patient unable to conceive
* receive the administration of a product that will interfere with the application of LABS™ Adhesion Barrier Material,
* receive the use of an approved or unapproved product or strategy for the purpose of preventing adhesion development,
* receive fibrin glue, surgical sealant, or other haemostatic agent,
* undergo an open procedure
* undergo a posterior colpotomy,
* undergo insufflation with a gas other than CO2,
* undergo Laprolift or similar device for elevation of the abdominal wall, as an alternative to CO2 insufflation,
* undergo abdominal cavity humidification or oxygenation,
* undergo robotic surgery,
* receive irrigants containing, glucocorticoids, antihistamines, heparin or antiseptic additives.
* have a postoperative drain
* does not have complete lysis of any adhesions to the posterior uterus
* has deep infiltrating endometriosis that is not treated during surgery
* patient had ovarian cysts with no other pathology
* be considered to have no clinical indication for a SLL

For the myomectomy sub study the patient:

* does not undergo laparoscopic myomectomy with at least (1) posterior uterine serosal incision of > 3 cm in length,
* has only pedunculated fibroids removed from the posterior aspect of the uterus
* has adenomyoma alone without fibroids
* has therapeutic hysteroscopy with treatment of congenital malformation, myomectomy or treatment of Asherman's syndrome
* excepting diagnostic hysteroscopy or polypectomy with lactated Ringer's solution (LRS) undertaken prior to laparoscopy and all fluid removed prior to laparoscopic filming.

Ages: 18 Years to 46 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2014-06 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events, abnormal changes in vital signs and/or clinical laboratory measures | Between baseline initial surgery and second look laparoscopy (4-12 weeks)

SECONDARY OUTCOMES:
Surgeon satisfaction with the device and it's application | During baseline initial surgery

OTHER OUTCOMES:
Patients with myomectomy | Baseline initial surgery to second look laparoscopy (4-12 weeks)
  Assessment in the change in adhesion score at the posterior uterus in the LABS™ treated patients compared to the surgery only controls.
Change in adhesion score of patients with other gynecological pathology | Baseline initial surgery to second look laparoscopy (4-12 weeks)
  Assessment of the change in adhesion score at sites of surgery in the LABS™ treated patients compared to the surgery only controls.
Other adhesion parameters | Baseline initial surgery to second look laparoscopy (4-12 weeks)
  The incidence of patients with adhesions; the number of pre-specified sites with adhesions, and the severity and extent of adhesions at these pre-specified anatomical locations.

CONTACTS AND LOCATIONS:
Overall Officials: Rudy DeWilde, MD, ScD, PhD, Principal Investigator — Professor and Head Department of Gynecology, Obstetrics and Gynecology Oncology, Pius-Hospital; Sara Y Brucker, MD, PhD, Principal Investigator — Deputy Head of Department of Gynecology and Obstetrics, University of Tubingen Women's Hospital; Matthias Korell, MD, Principal Investigator — Head Department of Obstetrics and Gynecology, Johanna Etienne-Krankenhaus; George A Pistofidis, MD, Principal Investigator — Director Department of Gynaecological Surgery Lefkos, Stavros Hospital; Geoffery H Trew, M.B.B.S, Study Director — Consultant in Reproductive Medicine and Surgery, Hammersmith Hospital
Locations (4):
- Germany (3):
  - Johanna Etienne Krankenhaus, Neuss
  - Pius-Hosptial, European Medical School Oldenburg-Groningen, Carl von Ossietzky University, Oldenburg
  - University of Tubingen Women's Hosptial, Tübingen
- Lefkos Stavros Hospital, Athens, Greece